CLINICAL TRIAL: NCT02168179
Title: Safety of Treatment With KeraStat Skin Therapy in Breast Cancer Patients Developing Radiation Dermatitis
Brief Title: KeraStat Skin Therapy in Treating Radiation Dermatitis in Patients With Newly Diagnosed Stage 0-IIIA Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer pursuing study at our site.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00028009; NCI-2014-01274 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 98114; P30CA012197 (NIH)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Ductal Breast Carcinoma in Situ; Skin Reactions Secondary to Radiation Therapy; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (KeraStat Skin Therapy) (Experimental): Patients apply KeraStat Skin Therapy topically BID during radiation therapy.
  Interventions: Procedure: dermatologic complications management/prevention; Other: questionnaire administration

INTERVENTIONS:
Procedure: dermatologic complications management/prevention — Apply KeraStat Skin Therapy topically
  Other Names: complications management/prevention, dermatologic; management/prevention, dermatologic complications
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies KeraStat Skin Therapy in treating radiation dermatitis in patients with newly diagnosed stage 0-IIIA breast cancer. Radiation dermatitis is an itchy, painful skin rash that can occur following treatment with radiation. KeraStat Skin Therapy may be a better treatment for radiation dermatitis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain a preliminary estimate the incidence of early adverse skin reaction (EASR) during radiation therapy (RT) and up to two months post RT after the application of the cosmetic cream KeraStat Skin Therapy during RT in breast cancer patients in a pilot study.

SECONDARY OBJECTIVES:

I. To associate personal characteristics (e.g., race/ethnicity, age, hormone therapy, smoking status, comorbidities, breast size) and treatment characteristics (e.g., RT dose) to incidence of EASR at any time point.

OUTLINE:

Patients apply KeraStat Skin Therapy topically twice daily (BID) during radiation therapy.

After completion of study treatment, patients are followed up at 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with breast carcinoma, stage 0-IIIA (including ductal carcinoma in situ [DCIS])
* Status post-lumpectomy, -quadrantectomy, or -mastectomy
* Plan to receive adjuvant radiation to the whole breast or chest wall +/- regional lymph nodes
* Total dose >= 40Gy
* Dose per fraction >= 1.8 use of 2-dimensional (2D), 3-dimensional (3D) conformal, or intensity-modulated radiation therapy (IMRT) treatment techniques allowed; skin sparing IMRT patients excluded; a daily fraction of 2.7 Gy to the whole breast is suggested for hypofractionated regimens
* Concurrent and sequential boost techniques are allowed for both standard and hypofractionated regimens
* Adjuvant hormonal therapy will be allowed prior to, during and/or after RT at the discretion of a medical oncologist
* Targeted therapies such as Herceptin will be allowed prior to, during, and/or after RT at the discretion of the medical oncologist
* Patients who are able and willing to sign protocol consent form

Exclusion Criteria:

* Prior radiation to the involved breast or chest wall
* Concurrent chemotherapy; (patients may receive chemotherapy prior to radiation or following radiation at the treating physician's discretion)
* Patients who underwent breast reconstruction following mastectomy (placement of tissue expanders and implants are not allowed)
* Patients undergoing partial breast irradiation
* Patients who have undergone MammoSite® or any other form of brachytherapy
* Patients may not be concurrently enrolled in a protocol that involves treatment of the skin ie: applying lotions /moisturizers; protocols that do not involve treatment of the skin are allowed
* Patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of any RT-induced EASR defined as a grade 4 or higher toxicity using the Modified Oncology Nursing Society Criteria for Radiation-Induced Acute Skin Toxicity | Up to 2 months after completion of radiation therapy
  At each time point the proportion of women who have RT-induced EASR present will be estimated and a 95% confidence interval will be calculated around this estimate.

OTHER OUTCOMES:
Categorical confounders, such as race/ethnicity, age, hormone therapy, smoking history/status, diabetes, high blood pressure, breast size, RT characteristics, and RT dosimetry characteristics, using the Baseline Study Risk Questionnaire | Baseline
  A series of 2xr tables will be examined to determine the relationship between each of the categorical confounders and the primary endpoint. Chi-squared statistics will be estimated for each of these tables to give some preliminary descriptive data to identify potential variables that may be associated with the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Blackstock, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States